CLINICAL TRIAL: NCT06717009
Title: A Prospective, Multicenter, Randomized Controlled Study of Three-dimensional Visualization Techniques to Improve the Quality and Safety of Robot-assisted Nephron Sparing Surgery for Complex Renal Tumors
Brief Title: A Study of 3D Visualization Techniques to Improve the Quality and Safety of Robot-assisted Nephron Sparing Surgery for Complex Renal Tumors.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking University First Hospital (Other); Liaoning Cancer Hospital & Institute (Other); The Second Affiliated Hospital of Dalian Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Qilu Hospital of Shandong University (Other); Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other); Hebei Medical University Fourth Hospital (Other); West China Hospital (Other); Tongji Hospital (Other); Sun Yat-sen University Tumor Hospital (Unknown); Shanghai Cancer Hospital, China (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E20241351
Record Dates: First submitted 2024-11-24; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Kidney Neoplasms / Surgery; Robotic Surgical Procedures; Imaging, Three-Dimensional / Methods; Nephrectomy / Methods
Keywords: Three-dimensional visualization technique;; Three-dimensional reconstruction; Robotic surgery; Kidney neoplasms; Laparoscopy; Nephron sparing surgery
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: The researchers will randomize participants into a 3D trial group and a conventional group for comparison. The 3D trials group will undergo preoperative 3D reconstruction, while the conventional group will only undergo routine CT/MRI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3D trial group (Experimental): The three-dimensional reconstruction data of patients will be synthesized according to renal enhanced CT/MRI within 48 hours before surgery. The surgeon/researcher will conduct surgical planning according to the results of the three-dimensional reconstruction and perform robot-assisted laparoscopic nephron sparing surgery.
  Interventions: Diagnostic Test: Preoperative three-dimensional reconstruction
- Conventional group (No Intervention): The patients will not undergo preoperative 3D reconstruction. The surgeon will arrange robot-assisted laparoscopic nephron sparing surgery according to routine CT/MRI.

INTERVENTIONS:
Diagnostic Test: Preoperative three-dimensional reconstruction — On the basis of conventional CT/MRI, the patient will undergo 3D reconstruction within 48 hours before surgery. The surgeon/researcher will conduct surgical planning according to the results of the 3D reconstruction and perform robot-assisted laparoscopic nephron sparing surgery.
  Arms: 3D trial group

SUMMARY:
The goal of this clinical trial is to learn the evidence-based medical value of 3D visualization techniques to improve tumor control, preservation of renal function, and perioperative safety in robot-assisted nephron sparing surgery for complex renal tumors. The main question it aims to answer is:

Is 3D visualization techniques more effective in improving robot-assisted nephron sparing surgery for complex renal tumors in terms of tumor control, renal function preservation, and perioperative safety.

The researchers will randomize participants into a 3D trial group and a conventional group for comparison.

Participants will:

Complete Blood routine, liver and kidney function tests on the first and third day after operation.

Have Renography at 3 and 12 months after the operation. Cooperate with follow-up visits.

DETAILED DESCRIPTION:
1. Sample size:

   When designing this experiment, considering the warm ischemic time reported by our center and in the literature, with a test power of 80% (β= 0.2), a power value of 0.8, a one-sided type I error of 2.5% (α= 0.05), the sample size is calculated to be 242 cases. The enrollment is planned to last 2 years, and the follow-up results from enrollment to the initial stage are for 5 years. Calculated based on a 30% dropout rate, 350 cases are planned to be enrolled.
2. Enrollment screening:

   Appropriate, reproducible methods should be used to evaluate the tumor prior to randomization (e.g., CT and/or MRI). The following evaluations should be made prior to randomization: demographic data, medical history (including concomitant disease and treatments), physical examination, pregnancy test (if necessary), special examinations (chest X-ray and ECG).

   The following evaluations should be made prior to randomization: vital signs and physical examination (including Karnofsky performance status score, height, and weight), hematological and biochemical examinations.
3. Randomization:

   Patients who meet the selection criteria will be randomly allocated to the 3D trial group and the conventional group in a 1:1 ratio.
4. Assessment During the Study Period:

   During the study period, patients' concomitant disease and treatments will be continuously monitored, and vital signs, weight, Karnofsky performance status score, hematological examinations (including white blood cells/neutrophils), and serum biochemical examinations will be conducted according to specified time intervals for each patient. An conventional ECG and chest X-ray/CT examination will be conducted prior to surgery. Tumor assessment will be conducted during the perioperative period (clinical examination, chest X-ray or chest CT/MRI, and abdominal CT/MRI). Laboratory examination indicators during the perioperative period should be recorded, such as preoperative and postoperative hematological and biochemical examinations. The focus is to complete the renogram to evaluate renal function within 1 month prior to surgery, and re-evaluating renal function with a renogram 3 months and 12 months after surgery to assess changes in renal function. No matter what surgical method is used, detailed records should be made of what was seen during the operation, the surgical method, operative data, and postoperative pathology. All patients should be followed up according to the study protocol, and PFS and OS should be recorded.
5. Statistical Analysis:

Statistical analysis will be conducted using the SPSS 24.0 software package. Statistical descriptions will use rates for enumeration data, and means and 95% confidence intervals for measurement data. The t-test will be used to compare the measurement data between the two groups, the Chi-square test will be used to analyze the enumeration data, the Kaplan-Meier method will be used to calculate the survival curve, and the Log-rank test will be used to compare the two treatments.HR and 95% Confidence intervals for survival in subgroups will be determined with the multiple individual Cox models, which will separately measure the interaction between factors and treatment effect. The probability P value will be used for statistical inference regardless of the stage, and the statistically significant difference thresholds will be adopted as 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. The imaging diagnosis is single renal cell carcinoma, clinical stage is T1N0M0-T2N0M0, and the contralateral kidney function is good.
2. Physical status and organ function allow robotic-assisted partial nephrectomy.
3. Be able to adhere to the protocol during the study.
4. The age ranges from 18 to 75 years, and there is no chronic kidney disease.
5. KPS > 80; ECOG score: 0-1; There are no other serious concomitant diseases and the organ function is good.
6. There are no medical contraindications seriously affecting anesthesia and surgery.
7. The patient has no history of other malignant tumors in the past 5 years.
8. There is no surgical history of epigastrium and the affected kidney.
9. Estimated survival is more than 6 months, and there are no other severe diseases that reduce survival to less than 5 years.

Exclusion Criteria:

1. Women who are pregnant or lactating, or who are of reproductive age and are not using effective contraception.
2. Comorbid serious medical diseases or conditions, for example, clinically severe or active heart disease, severe uncontrolled medical illnesses and infections, severe uncontrolled digestive disorder, severe electrolyte disturbance, active disseminated intravascular coagulation, major organ failure such as decompensated cardiac, pulmonary, hepatic, or renal failure, symptomatic peripheral neuropathy. Can not tolerate robot-assisted laparoscopic partial nephrectomy
3. Organ transplant recipients requiring immunosuppressive therapy.
4. There is history of other malignancies within 5 years of trial initiation, excluding cured basal cell carcinoma of the skin and carcinoma in situ of the cervix.
5. Patients who have received biological therapy or other anticancer traditional Chinese medicine within 4 weeks.
6. Patients with multiple or bilateral renal tumors or solitary renal tumors.
7. Patient without complete clinical information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
warm ischemia time | From start of arterial clamping to release of arterial blocking forceps during surgery, an average of 25 minutes.
  The time from start of arterial clamping to release of arterial blocking forceps during surgery. Superselective arterial blockade will be recorded separately as a specific blockade modality. The arterial blocking time will be recorded as 0 for those without arterial blockage.

SECONDARY OUTCOMES:
operative time | From the beginning to the end of the surgery, an average of 3 hours.
Intraoperative bleeding | From the beginning to the end of the surgery, an average of 3 hours.
Length of postoperative hospital stay | an average of a week.
Incidence of postoperative complications | an average of a week.
Positive rate of pathological margin | an average of a week.
Conversion rate | From the beginning to the end of the surgery, an average of 3 hours.
  Laparoscopic surgery converts to open surgery, or partial nephrectomy converts to radical nephrectomy during the surgery.
Postoperative creatinine changes | 1 month
Changes in glomerular filtration rate | 3 month.
3-year recurrence-free survival rate | Within three years from the end of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen XS, Zhang ZT, Du J, Bi XC, Sun G, Yao X. Optimal surgical margin in nephron-sparing surgery for T1b renal cell carcinoma. Urology. 2012 Apr;79(4):836-9. doi: 10.1016/j.urology.2011.11.023. Epub 2012 Feb 2. PMID 22305422
- [Background] Piramide F, Kowalewski KF, Cacciamani G, Rivero Belenchon I, Taratkin M, Carbonara U, Marchioni M, De Groote R, Knipper S, Pecoraro A, Turri F, Dell'Oglio P, Puliatti S, Amparore D, Volpi G, Campi R, Larcher A, Mottrie A, Breda A, Minervini A, Ghazi A, Dasgupta P, Gozen A, Autorino R, Fiori C, Di Dio M, Gomez Rivas J, Porpiglia F, Checcucci E; European Association of Urology Young Academic Urologists and the European Section of Uro-Technology. Three-dimensional Model-assisted Minimally Invasive Partial Nephrectomy: A Systematic Review with Meta-analysis of Comparative Studies. Eur Urol Oncol. 2022 Dec;5(6):640-650. doi: 10.1016/j.euo.2022.09.003. Epub 2022 Oct 7. PMID 36216739
- [Background] Amparore D, Pecoraro A, Checcucci E, Piramide F, Verri P, De Cillis S, Granato S, Angusti T, Solitro F, Veltri A, Fiori C, Porpiglia F. Three-dimensional Virtual Models' Assistance During Minimally Invasive Partial Nephrectomy Minimizes the Impairment of Kidney Function. Eur Urol Oncol. 2022 Feb;5(1):104-108. doi: 10.1016/j.euo.2021.04.001. Epub 2021 Apr 24. PMID 33903083
- [Background] Porpiglia F, Fiori C, Checcucci E, Amparore D, Bertolo R. Hyperaccuracy Three-dimensional Reconstruction Is Able to Maximize the Efficacy of Selective Clamping During Robot-assisted Partial Nephrectomy for Complex Renal Masses. Eur Urol. 2018 Nov;74(5):651-660. doi: 10.1016/j.eururo.2017.12.027. Epub 2018 Jan 6. PMID 29317081
- [Background] Gu L, Liu K, Du S, Li H, Ma X, Huang Q, Ai Q, Chen W, Gao Y, Fan Y, Xie Y, Yao Y, Wang H, Li P, Xuan Y, Wang B, Zhang X. Prediction of pentafecta achievement following laparoscopic partial nephrectomy: Implications for robot-assisted surgery candidates. Surg Oncol. 2020 Jun;33:32-37. doi: 10.1016/j.suronc.2020.01.004. Epub 2020 Jan 7. PMID 32561096
- [Background] Sagalovich D, Dagenais J, Bertolo R, Garisto JD, Kaouk JH. Trifecta Outcomes in Renal Hilar Tumors: A Comparison Between Robotic and Open Partial Nephrectomy. J Endourol. 2018 Sep 12;32(9):831-836. doi: 10.1089/end.2018.0445. PMID 29984597
- [Background] Cacciamani GE, Medina LG, Gill T, Abreu A, Sotelo R, Artibani W, Gill IS. Impact of Surgical Factors on Robotic Partial Nephrectomy Outcomes: Comprehensive Systematic Review and Meta-Analysis. J Urol. 2018 Aug;200(2):258-274. doi: 10.1016/j.juro.2017.12.086. Epub 2018 Mar 24. PMID 29580709
- [Background] Weight CJ, Larson BT, Fergany AF, Gao T, Lane BR, Campbell SC, Kaouk JH, Klein EA, Novick AC. Nephrectomy induced chronic renal insufficiency is associated with increased risk of cardiovascular death and death from any cause in patients with localized cT1b renal masses. J Urol. 2010 Apr;183(4):1317-23. doi: 10.1016/j.juro.2009.12.030. Epub 2010 Feb 19. PMID 20171688